CLINICAL TRIAL: NCT04988386
Title: An Open-Label Extension and Safety Monitoring Study of Acoramidis (AG10) in Participants With Symptomatic Transthyretin Amyloid Cardiomyopathy Who Completed the Phase 3 ATTRibute-CM Trial (AG10-301)
Brief Title: Open-Label Safety Study of Acoramidis (AG10) in Symptomatic ATTR Participants
Acronym: AG10
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eidos Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG10-304; 2020-005643-22 (EudraCT Number)
Record Dates: First submitted 2021-07-13; First posted 2021-08-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Amyloid Cardiomyopathy, Transthyretin-Related
Keywords: ATTR-CM
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — attruby

STUDY DESIGN:
Intervention Model Description: Open-label study extension study from the AG10-301 double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AG10 (Experimental): Open-label study all participants will receive AG10 during this study.
  Interventions: Drug: Acoramidis (AG10)

INTERVENTIONS:
Drug: Acoramidis (AG10) — Acoramidis (AG10) twice daily
  Other Names: AG10; ALXN 2060

SUMMARY:
Open-Label Extension and Safety Monitoring Study of Acoramidis (AG10) in Participants with Symptomatic Transthyretin Amyloid Cardiomyopathy Who Completed the Phase 3 ATTRibute-CM Trial (AG10-301)

DETAILED DESCRIPTION:
The primary objective of this prospective, multi-center, open-label study is to evaluate the long-term safety and tolerability of acoramidis in patients with an established diagnosis of ATTR-CM and heart failure who are concomitantly treated with currently recommended heart failure therapies. Secondary efficacy and PD objectives will be assessed. Exploratory objectives may also be assessed.

All participants who complete 30 months of blinded study treatment and the Month 30 assessments of the double-blind treatment period of the Phase 3 ATTRibute-CM trial (AG10-301) may be eligible to participate in this Open Label Extension (OLE) study of acoramidis. The Day 1 visit in Study AG10-304 may be the same as the Month 30 visit in Study AG10-301. Under these circumstances, the last dose of Investigational Medicinal Product (IMP) in Study AG10-301 (either blinded acoramidis or matching placebo) will be the night before the day of the Month 30 visit. The first dose of open-label acoramidis in Study AG10-304 will be during the Study AG10-304 Day 1 visit after baseline assessments have been completed.

Currently, tafamidis is approved for the treatment of ATTR-CM in some regions. Participants are not allowed to be treated with tafamidis or any other ATTR-CM-specific approved or investigational treatment, or therapies used off-label or as non-prescription supplements for ATTR-CM at any time during the study. If participants choose treatment with an alternative treatment as described above, they will be asked to discontinue acoramidis and complete an End of Treatment (EoT) form, and they may be asked to discontinue/withdraw from the study. If a participant discontinues/withdraws from the study, the participant will be asked to complete an early termination visit and a safety follow-up visit.

Participants are not permitted to participate in another interventional clinical trial (except Study AG10-301) within 30 days prior to dosing and throughout Study AG10-304. Participants who choose to participate in another interventional clinical trial will be asked to withdraw from acoramidis and complete an EoT form, and they may be asked to discontinue/withdraw from the study. If a participant discontinues/withdraws from the study, the participant will be asked to complete an early termination visit and a safety follow-up visit. Participation in observational and/or registry studies should be discussed with the Medical Monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Completed 30 months of the blinded study treatment in Study AG10-301 and the Study AG10-301 Month 30 visit including assessments and procedures.
2. Have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.
3. Female participants of childbearing potential who engage in heterosexual intercourse must agree to use a highly effective method of contraception beginning with enrollment and continuing for 30 days after the last dose of acoramidis. Female participants using oral contraceptives must agree to use an additional birth control method. While not considered highly effective, a double-barrier method is acceptable. A male participant who is sexually active with a female of childbearing potential and has not had a vasectomy must agree to use a double-barrier method of birth control.

Exclusion Criteria:

1. Acute myocardial infarction, acute coronary syndrome or coronary revascularization within 90 days prior to Day 1 stroke or transient ischemic attack (TIA) within 90 days prior to Day 1.
2. Has hemodynamic instability, that in the judgment of the Investigator, would pose too great a risk for participation in the study.
3. Has had a heart and/or liver transplant or is on the heart transplantation list within the year prior to Day 1
4. Has had implantation of a cardiac mechanical assist device (CMAD) or is scheduled for implantation of a CMAD
5. Has confirmed diagnosis of light-chain (AL) amyloidosis at any time during Study AG10-301.
6. Has estimated glomerular filtration rate (eGFR) by modification of diet for renal disease (MDRD) formula < 15 mL/min/1.73 m2 at Month 27 of Study AG10-301 or at any subsequent central lab value prior to Day 1.
7. Known hypersensitivity to acoramidis, its metabolites, or formulation excipients.
8. At the end of Study AG10-301 or at Day 1 of Study AG10-304 (or any time during the study), participant is on prohibited medication.
9. Females who are pregnant or breastfeeding. A negative urine pregnancy test at the Day 1 visit and at each study visit are required for female participants of childbearing potential.
10. In the judgment of the Investigator or Medical Monitor, has any clinically important ongoing medical condition or laboratory abnormality or condition that might jeopardize the participant's safety, increase their risk from participation, or interfere with the study.
11. Participation in another interventional clinical trial (with the exception of Study AG10-301) within 30 days prior to dosing. Participation in observational and/or registry studies should be discussed with the Medical Monitor.
12. Has any condition that in the opinion of the Investigator or Medical Monitor would preclude compliance with the study protocol such as a history of substance abuse, alcoholism, or a psychiatric condition.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2028-04-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent Adverse Events [Safety and Tolerability] | 60 months
  Incidence of each treatment-emergent adverse events measured over 60 Months or study completion

SECONDARY OUTCOMES:
Evaluate all-cause mortality and cardiovascular mortality | 60 months
  Assessment of All-cause mortality and CV mortality during study period
Evaluate the effect of acoramidis on the 6-minute walk test (6MWT) | 60 months
  Change from Baseline in distance walked during the 6MWT during study period
Evaluate the effect of acoramidis on health-related quality of life Kansas City Cardiomyopathy Questionnaire | 60 months
  Change from Baseline in Kansas City Cardiomyopathy Questionnaire Overall Score during study period [scale is scored from 0-100, where 0=Poor, 100=Excellent]
Evaluate the effect of acoramidis on the frequency of CV-related hospitalization | 60 months
  assess CV-related hospitalization during the study period

CONTACTS AND LOCATIONS:
Locations (72):
- United States (26):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado Hospital - Anschutz Medical Campus, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - MedStar Medical Group Cardiology at Franklin Square, Baltimore, Maryland
  - Boston University Medical Center General Clinical Research Unit, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - New York University Langone Health, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Laurelton Heart Specialists, Rosedale, New York
  - Montefiore Medical Center at Hutchinson, The Bronx, New York
  - Duke University Health System - Duke Clinic, Durham, North Carolina
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Roanoke Heart Institute, Roanoke, Virginia
  - University of Washington School of Medicine, Seattle, Washington
  - Providence Sacred Heart Children's Hospital, Spokane, Washington
- Australia (6):
  - Saint Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende - Campus Sint-Jan, Bruges, West Vlaanderen
- Brazil (3):
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Centro Avançado de Pesquisa e Estudos para o Diagnóstico CAPED, Ribeirão Preto, São Paulo
  - Instituto do Coração de São Paulo, São Paulo, São Paulo
- Canada (8):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Saint Boniface Hospital, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre - Halifax Infirmary, Halifax, Nova Scotia
  - Toronto Heart Centre, Toronto, Ontario
  - L' Institut de Cardiologie de Montréal, Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Hôpital régional de Rimouski, Rimouski, Quebec
- Czechia (3):
  - Vseobecna Fakultni Nemocnice v Praze, Prague, Prague
  - Institut Klinické a Experimentální Medicíny, Prague, Prague
  - Fakultní Nemocnice u sv. Anny v Brně, Brno, South Moravian
- Aarhus Universitets Hospital, Aarhus N, Palle Juul-Jensens, Denmark
- Alexandra General Hospital of Athens, Athens, Attica, Greece
- Mater Misericordiae University Hospital, Dublin, Dublin, Ireland
- Israel (2):
  - The Chaim Sheba Medical Center, Ramat Gan, Tel Aviv
  - Hadassah University Hospital Ein Kerem, Jerusalem
- Italy (4):
  - Ospedale San Donato, Arezzo, Arezzo
  - Azienda Ospedaliero - Universitaria Careggi, Florence, Florence
  - Fondazione Toscana Gabriele Monasterio per la Ricerca Medica e di Sanità Pubblica, Pisa, Pisa
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen, Provincie Groningen
  - Universitair Medisch Centrum Utrecht, Utrecht, Utrecht
- New Zealand (2):
  - Middlemore Clinical Trials - Middlemore Hospital, Papatoetoe, Auckland
  - Waikato Hospital, Hamilton, Waikato Region
- Centro Hospitalar Universitário Lisboa Norte EPE- Hospital Santa Maria, Lisbon, Lisbon District, Portugal
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Gyeonggi-do
- Spain (6):
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, La Coruña
  - Clinica Universidad de Navarra Madrid, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
- United Kingdom (2):
  - National Amyloidosis Centre, Division of Medicine - Royal Free, London, England
  - Richmond Pharmacology Ltd, London, England

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alexander KM, Davis MK, Akinboboye O, Berk J, Bhatt K, Cappelli F, Cuddy SAM, Fontana M, Garcia-Pavia P, Gillmore JD, Griffin JM, Grodin JL, Judge DP, Khouri MG, Lam K, Masri A, Maurer MS, Obici L, Ruberg FL, Sarswat N, Shah K, Soman P, Stern L, Wright R, Xiong K, Cao X, Lystig T, Tamby JF, Castano A, Katz L, Sinha U, Fox JC, Solomon SD, Grogan M. Efficacy of Acoramidis in Wild-Type and Variant Transthyretin Amyloid Cardiomyopathy: Results From ATTRibute-CM and Its Open-Label Extension. JAMA Cardiol. 2026 Jan 1;11(1):57-67. doi: 10.1001/jamacardio.2025.4477. PMID 41205147
- [Derived] Judge DP, Gillmore JD, Alexander KM, Ambardekar AV, Cappelli F, Fontana M, Garcia-Pavia P, Grodin JL, Grogan M, Hanna M, Masri A, Nativi-Nicolau J, Obici L, Hvitfeldt Poulsen S, Sarswat N, Shah K, Soman P, Lystig T, Cao X, Wang K, Pecoraro ML, Tamby JF, Katz L, Sinha U, Fox JC, Maurer MS. Long-Term Efficacy and Safety of Acoramidis in ATTR-CM: Initial Report From the Open-Label Extension of the ATTRibute-CM Trial. Circulation. 2025 Mar 4;151(9):601-611. doi: 10.1161/CIRCULATIONAHA.124.072771. Epub 2024 Nov 18. PMID 39556242